CLINICAL TRIAL: NCT02825381
Title: Evaluation of Routine One-Stage Exchange Procedure for Chronically Infected Total Hip Arthroplasty
Brief Title: One-Stage Exchange for Chronically Infected Total Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-46
Record Dates: First submitted 2014-01-08; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-01

CONDITIONS: Infection
Keywords: Arthroplasty; Hip
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary goal of the study is to evaluate the success rate of routine one-stage exchange for treatment of chronically infected total hip arthroplasty performed at the investigators institution, and to compare it to the current literature reporting success rate of selected one-stage exchange procedure or two-stage procedure.

The secondary goal is to detect the potential prognostic factors and potential selection criteria which may influence the success rate. The tested hypothesis is following: the success rate of routine one-stage exchange is lower than that of selected one-stage or two-stage procedure

ELIGIBILITY:
Inclusion Criteria:

* Chronically infected total hip Arthroplasty
* One-stage exchange procedure operated on at the investigators institution between January 1, 2007 and November 30, 2010

Exclusion Criteria:

* Patient refused to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases operated on at the investigators institution between January 1, 2007 and November 30, 2010
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
infection of the prosthesis | For the duration of hospital stay, up to 1 year]
  Rate of diagnosis infection of the prosthesis

CONTACTS AND LOCATIONS:
Locations (1):
- CCOM, Hôpitaux Universitaires de Strasbourg, Illkirch-Graffenstaden, Bas Rhin, France